CLINICAL TRIAL: NCT01555333
Title: An Open-Label Extension Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in Subject With Fragile X Syndrome
Brief Title: An Open Label Extension Study in Subjects With Fragile X Syndrome
Acronym: 209FX303
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209FX303
Record Dates: First submitted 2012-03-01; First posted 2012-03-15 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — arbaclofen placarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arbaclofen (Experimental): Open Label Study
  Interventions: Drug: arbaclofen

INTERVENTIONS:
Drug: arbaclofen — A flexible dose titration will be utilized. Orally disintegrating tablets
  Other Names: STX209

SUMMARY:
This study will enroll subjects who have completed Protocols 209FX301, 209FX302, or are currently participating in Protocol 2202 into a long-term study in which all subjects will receive active drug (arbaclofen).

DETAILED DESCRIPTION:
Three studies sponsored by Seaside Therapeutics, Inc., are currently evaluating the efficacy of STX209 for management of typical problem behaviors in subjects with FXS. These are Study 209FX301, "A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of STX209 (Arbaclofen) Administered for the Treatment of Social Withdrawal in Adolescents and Adults with Fragile X Syndrome;" Study 209FX302, "A Randomized, Double-Blind, Placebo-Controlled, Fixed- Dose Study of the Efficacy, Safety, and Tolerability of STX209 (Arbaclofen) Administered for the Treatment of Social Withdrawal in Children with Fragile X Syndrome;" and Study 22002, "An Open-Label Extension Study to Evaluate the Safety, Tolerability and Pharmacokinetics of STX209 in Subjects with Fragile X Syndrome." This study will enroll subjects who have completed Protocols 209FX301, 209FX302, or are currently participating in Protocol 22002 into a long-term, open-label study. The open-label extension protocol will provide data on the long-term safety and tolerability of STX209 among subjects with FXS who receive treatment under conditions reflective of their typical medical care rather than in their previously completed study.

ELIGIBILITY:
Inclusion Criteria:

1. Successfully completed all scheduled visits of the previous protocol ( 22002, 209FX301, or 209FX302).
2. A parent,LAR, or caregiver must be willing and able to accompany the subject to all study visits, participate in phone calls, complete study assessments, administer study medication, and report the subject's condition and medication use to site staff members.
3. Prior to the conduct of any study-specific procedures, the subject must provide written informed consent to participate in the study ( if developmentally appropriate) or verbal assent and the parent/caregiver/LAR must provide written informed consent. If the caregiver attending the clinic visits is not the parents, caregiver, or LAR, written consent must also be obtained for the caregiver's participation in the study.
4. Current treatment with no more than 3 psychoactive medications, including anti-epileptics, unless the Medical Monitor is consulted.
5. Subjects with a history of seizure disorder must have been seizure free for 6 months and be taking anti-epileptics, or seizure free for 3 years if not receiving anti-epileptic treatment. If currently receiving treatment with anti-epileptics, serum concentration levels must be tested and be in therapeutic range.
6. Negative pregnancy test for females of childbearing potential or be using a medically acceptable form of birth control.

Exclusion Criteria

1. Subjects with any condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. This includes, but is not limited to impairment of renal function, evidence or history of malignancy or any significant hematological, endocrine, cardiovascular, respiratory, hepatic, or gastrointestinal disease.
2. Subjects who are currently engaged in illicit drug or alcohol abuse.
3. Subjects who had a serious adverse event (SAE) while taking STX209 during their previous protocol (22002,209FX301,309FX302)that the Investigator considered related to STX209, unless approval from the Medical Monitor is obtained.
4. The occurrence or continuation of any AE or condition during Studies 22002, 209FX301, or 209FX302 that, in the opinion of the Investigator, should exclude this subject from participating in the open-label extension.
5. Subjects taking another investigational drug, other than STX209, currently or within 30 days of Visit 1. Subject must not take any investigational drugs during this study.
6. Subjects who, in the Investigator's opinion, might not be suitable for the study.
7. Subjects treated with vigabatrin, tiagabine, or riluzole currently or within 2 weeks of Visit 1.
8. Subjects treated with racemic baclofen currently or within 1 week of Visit 1.

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 357 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety Measures | 100 weeks
  Adverse Events, Suicidality Assessment, Physical Examination, Vital Signs and Weight, Laboratory Tests: Complete Blood Count, Urinalysis, Chemistry Panel

SECONDARY OUTCOMES:
Efficacy | 100 Weeks
  Aberrant Behavior Checklist Lethargy/Social Withdrawal Sub- Scale Clinical Global Impression Vineland Adaptive Behavior Scales Stanford Binet Intelligence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, M.D., Study Director — Seaside Therapeutics, Inc.
Locations (23):
- United States (23):
  - Seaside Therapeutics Site #16, Phoenix, Arizona
  - Seaside Therapeutics Site #07, Long Beach, California
  - Seaside Therapeutics Site #10, Sacramento, California
  - Seaside Therapeutics Site #17, Aurora, Colorado
  - Seaside Therapeutics Site #01, Miami, Florida
  - Seaside Therapeutics Site #14, Orange City, Florida
  - Seaside Therapeutics Site #20, Decatur, Georgia
  - Seaside Therapeutics Site #02, Chicago, Illinois
  - Seaside Therapeutics Site #23, Kansas City, Kansas
  - Seaside Therapeutics Site #12, Baltimore, Maryland
  - Seaside Therapeutics Site #08, Worcester, Massachusetts
  - Seaside Therapeutics Site #03, Columbia, Missouri
  - Seaside Therapeutics Site #22, New York, New York
  - Seaside Therapeutics Site #04, Staten Island, New York
  - Seaside Therapeutics Site #24, Chapel Hill, North Carolina
  - Seaside Therapeutics Site #21, Durham, North Carolina
  - Seaside Therapeutics Site #05, Akron, Ohio
  - Seaside Therapeutics Site #15, Oklahoma City, Oklahoma
  - Seaside Therapeutics Site #11, Media, Pennsylvania
  - Seaside Therapeutics Site #19, Nashville, Tennessee
  - Seaside Therapeutics Site #25, Houston, Texas
  - Seaside Therapeutics Site #18, San Antonio, Texas
  - Seaside Therapeutics Site #13, Seattle, Washington